CLINICAL TRIAL: NCT04811534
Title: Qualitative Exploratory Study Among Reunionese Women and Their Partners Who Have a Child With Trisomy 21
Acronym: QUALI-21
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/06
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interview — Mixed exploratory study, mixing a mainly qualitative study (semi-directed interviews) with a descriptive observational study (short self-questionnaire of the interviewees).

SUMMARY:
According to data from French congenital malformation registries, the prevalence of Down Syndrome (DS) in 2017 (live births and medical termination of pregnancy (MToP)) in Reunion Island was the lowest in France (23.04 per 10,000 births), notably in relation to a young maternal age. However, if we look at live births, Reunion Island has the highest prevalence of DS in France (12.24 vs. 5.81 per 10,000 births), despite a well organized prenatal diagnosis (PND). In fact, the use of MToP in this context is the lowest in France (10.8 vs 26.3 per 10 000 births).

Local specificities may have an impact on the choice of patients to undergo or not undergo a MToP in the context of PND of DS and explain why the rate of recourse to MToP is the lowest in France. To date, no qualitative study exploring the reasons why women and their partners do not undergo a MToP in the context of DS has been conducted in Reunion Island.

Thus, the main hypothesis is that the low recourse to MToP following PND of DS in Reunion Island could be explained by the beliefs, values or choices of Reunion Island women and their partners during pregnancy in relation to a specific family, socio-cultural and economic context.

ELIGIBILITY:
Inclusion Criteria:

Parents:

* of a child born alive with Down Syndrome as of January 1, 2019 and registered within REMACOR
* living on the island of Reunion at the time of birth
* having a good understanding of French and/or Creole
* having given their written consent to the study

Exclusion Criteria:

Parents:

* with normal/negative prenatal screening (False positive)
* minors at the time of inclusion
* under guardianship or legal protection
* with a pathology preventing the interviews from taking place

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of a child born with Down Syndrome as of January 2019 living on the Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Reasons and motivations that lead parents living in Reunion Island not to carry out a medical termination of pregnancy, following a prenatal diagnosis of Down Syndrome | 1 day
  Collecting verbal data (verbatim) during individual semi-directive interviews with a French and Creole-speaking interviewer, trained in qualitative interviews with an audio recording, and then a written transcription of these verbatims. Women and their partners will be interviewed individually.
  The parents will be asked to recount chronologically the course of the pregnancy from the preconceptional period to the birth, focusing on their experiences during each stage of this period.
  Given the sensitivity of the subject, individual interviews are preferred to focus groups.

SECONDARY OUTCOMES:
Reasons that lead parents living in Reunion to carry out or not a prenatal diagnosis, among women who have had a child with Down Syndrome | 1 day
  Verbal data collection (verbatim) during individual semi-structured interviews of parents, by a French and Creole speaking interviewer, trained in qualitative interviews with an audio recording, followed by a written transcription of these verbatims. Women and their partners will be interviewed individually.
  For this criterion, the parents interviewed will be adults living in Reunion who have or have not wished to have a prenatal diagnosis of Down Syndrome for their child.
Socio-demographic characteristics of the parents and the pregnancy follow-up data of the women interviewed using a questionnaire and REMACOR data from the computerized medical record | 1 day
  Socio-demographic characteristics will be collected through a self-administered questionnaire, distributed after the individual qualitative interview. The questionnaire consists of 5 parts (socio-demographic data, health insurance, family, housing and religion) and 18 questions. The time required to complete the questionnaire is 10 minutes. This questionnaire will make it possible to describe the population surveyed on certain variables and to ensure that a reasoned sample (heterogeneous population) has been taken from the parents.

CONTACTS AND LOCATIONS:
Locations (2):
- Reunion (2):
  - CHU de la Réunion, Saint-Denis
  - CHU de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No